CLINICAL TRIAL: NCT00300157
Title: French Multicenter Study Assessing Angioplasty With Taxus Drug Eluting Stent in Unprotected Left Main Coronary Artery Associated to Other Coronary Lesions or Not
Brief Title: Left Main Coronary Artery Stenosis and Angioplasty With Taxus Stent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Didier Carrié, Rangueil Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-06
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Coronary Arteriosclerosis
Keywords: Left main coronary artery stenosis, stent, Taxus; Unprotected left main coronary artery disease; Percutaneous coronary intervention with Taxus stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Percutaneous coronary intervention with Taxus stent

SUMMARY:
The purpose of this study is to determine whether percutaneous coronary angioplasty with Taxus drug eluting stent is safe and effective in the treatment of unprotected left main coronary artery disease associated to other coronary lesions or not.

DETAILED DESCRIPTION:
Coronary artery bypass graft is the reference treatment of left main coronary artery disease. With the advancements of technology and particularly drug-eluting stents, in-stent restenosis has dramatically decreased and now it is possible to extend indications of complexes lesions such as left main coronary artery stenoses. In these particular situations,some centers performed percutaneous coronary angioplasty (PCI) with drug-eluting stents with acceptable results in terms of safety and efficacy. However, these procedures are performed at isolated sites and are not evaluated in multicenter trial.The aim of this study is to assess the safety and efficacy of this PCI with Taxus-stent in a french multicenter trial and to evaluate clinical and angiographic outcome of these patients at long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be > or = 18 years of age
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Ethics Committee
* Aspirin + Clopidogrel > or = 12 hours before percutaneous coronary intervention (PCI)
* Documented evidence of ischemic heart disease (clinical,biological or ECG) with unprotected left main coronary artery stenosis > or = 50% associated to other coronary lesions or not responsible of stable or unstable coronary syndrome above 48 hours
* The target reference vessel diameter must be > or = 2.5 mm
* Unprotected left main coronary artery disease eligible by coronary stenting

Exclusion Criteria:

* Restenosis lesion in left main coronary artery
* Known allergies to the following: aspirin, clopidogrel,ticlopidine,contrast agent or drug similar to paclitaxel
* Acute coronary syndrome < 48 hours
* Impaired renal function (creatinine > 180 ùmol/l) at the time of treatment
* Life expectancy less than 36 months
* Female of childbearing potential without reliable birth control
* Currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Coronarography | 9 months

SECONDARY OUTCOMES:
Major cardio-vascular events | 1, 18 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Didier Carrié, MD-PhD, Principal Investigator — Rangueil Hospital Toulouse France; Hélène ELTCHANINOFF, MD-PhD, Study Chair — Hôpital Charles Nicolle Rouen FRANCE; Thierry LEFEVRE, MD, Study Chair — Hôpital Jacques Cartier ICPS Massy FRANCE; Marc SILVESTRI, MD, Study Chair — Polyclinique du Parc Rambot Aix en Provence FRANCE
Locations (26):
- France (26):
  - Polyclinique du Parc Rambot, Aix-en-Provence
  - Clinique Rhône Durance, Avignon
  - Clinique Saint Augustin, Bordeaux
  - Chu Brest, Brest
  - CHU CAEN, Caen
  - Hôpital Cardiologique, Lille
  - Clinique du Tonkin, Lyon
  - Unité Cardio-Vasculaire, Marseille
  - CHU NORD, Marseille
  - Institut Hospitalier Jacques Cartier-ICPS, Massy
  - Hôpital Bon Secours, Metz
  - Clinique du Millénaire, Montpellier
  - Nouvelles Cliniques Nantaises, Nantes
  - Hôpital privé Les Franciscaines, Nîmes
  - CHU Caremeau, Nîmes
  - Hôpital COCHIN, Paris
  - Institut Mutualiste Montsouris, Paris
  - Groupe Hospitalier La Pitié-Salpetrière, Paris
  - CHU Pontchaillou, Rennes
  - Clinique Saint Hilaire, Rouen
  - Hôpital Charles Nicolle, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - Institut Arnaud Tzanck, Saint-Laurent-du-Var
  - CHU Toulouse Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - Clinique Saint Gatien, Tours